CLINICAL TRIAL: NCT02551081
Title: Genomic Sequencing and Personalized Treatment for Birth Defects in Neonatal Intensive Care Units
Status: Recruiting | Type: Observational
Sponsor: Children's Hospital of Fudan University (Other)
Collaborators: Xiamen Children's Hospital, Fujian of China (Other); Maternal and Child Health Hospital of Guangxi Zhuang Autonomous Region (Other); Guangzhou Women and Children's Medical Center (Other); Second Affiliated Hospital of Wenzhou Medical University (Other); Maternal and Child Health Hospital of Hubei Province (Other); The Maternal & Children Health Hospital of Dehong, Yunnan of China (Other)
Responsible Party: Sponsor
Other Study IDs: CHFudanU_NNICU2; NCT02607189 (obsolete NCT alias)
Record Dates: First submitted 2015-09-04; First posted 2015-09-16 (Estimated); Last update posted 2025-09-05 (Actual); Status verified 2025-09

CONDITIONS: Genetic Disease; Multiple Malformation; Congenital Malformation
MeSH Terms: conditions — Genetic Diseases, Inborn; Congenital Abnormalities

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Birth Defects: Neonates were diagnosed as birth defects who were recieving genomic sequencing and personalized treatment in NICU.

SUMMARY:
The purpose of study is to evaluate the benefits of using the Next Generation Sequencing Technology to diagnose birth defects and genetic diseases. The results from genomic sequencing can also significantly shorten the time of examination, improve the diagnosis rate, guide the clinical treatments. So the ultimate goal is individualized or personalized therapy and promote prognosis.

DETAILED DESCRIPTION:
Neonatal congenital malformation is one of the most frequent cause of infant death in the western world and major cities of China. There are many different types of congenital malformations, and some of these can be caused by changes in gene mutation. Next generation sequencing (NGS) is a high-throughput parallel sequencing that can provide genetic information with high accuracy. It is a faster and cost-effective method to detect gene mutations compared to Sanger sequencing. We hope to couple genomic techniques with more traditional methods involved in genetic discovery in order to investigate a broad range of conditions for which there is strong evidence that genetic factors are involved. So In this study, we evaluated the clinical role of NGS testing for neonatal genetic disease in newborns compared to Sanger sequencing to observe whether this new technology can significantly shorten the time of examination, improve the diagnosis rate, guide the intervention treatments and promote prognosis.

These neonates who have an undiagnosed illness, and partial families, will be eligible to participate in the study. The study population will be recruited from Children's Hospital of Fudan University inpatient population, primarily the neonatal intensive care unit (NICU), with a subpopulation presenting to other hospitals in China. All affected study participants will receive a genetic screening according to their clinical symptom. All subjects will have blood drawn for DNA isolation and genomic sequencing at the time of enrollment in the study. All blood sample volumes will adhere to the Fudan procedure on maximum blood in pediatric patients. In addition, cerebrospinal fluid and tissue samples may be collected and stored in the bank of biosamples. DNA will be isolated and prepared for NGS or Sanger with Fudan protocols at the Translational Medicine Center of Children's Hospital of Fudan University. Partial familial samples will also be obtained, and nucleic acids will also be sequenced, as indicated, to assist in diagnosis of the genetic disease in the newborn. All sequencing data will be stored in the Genome Center Biorepository. In the case of positive study findings that may be diagnostic, our investigator will perform confirmatory clinical diagnostic testing and, if confirmed, a standard clinical diagnostic report will be placed in the patient's medical record. Follow up with the patient's family will be guided by the clinical care team. Both molecular diagnoses results and duration to diagnosis will be recorded as primary outcomes.

In addition, this information will help alleviate anxiety on the part of the family, and also provides a mechanism for patient crossover into the rapid NGS arm if the patient is clinically deteriorating, and at the clinical care team's request. Each time a study participant is enrolled, the clinician and parents will be asked to fill out a survey prior to NGS testing and after return of results. We will also review the patient's medical record and collect clinical variables including laboratory testing, radiology results, medications and other treatments received to further analyze the effect NGS has on clinical care. So the ultimate goal is individualized or personalized therapy. We plan to follow up with families annually up to 18 months post enrollment and record clinical outcomes related to this study.

ELIGIBILITY:
Inclusion Criteria:

One of the following criteria required.

1. Neonates admitted to the Neonatal Intensive Care Units in one of the study hospitals
2. Clinical genetic testing or a genetic consult is ordered
3. Subject has one major structural anomaly or three or more minor anomalies
4. Abnormal laboratory testing suggestive of a genetic disease
5. Abnormal response to standard therapy for a major underlying condition

Exclusion Criteria:

1. Previously performed exome/genome sequencing on patient
2. Any infant in which clinical considerations preclude drawing 1.0 ml of blood
3. Has features pathognomonic for a large chromosomal aberration (Trisomy 13, 18, 21 or other)
4. Parents are unwilling to have genomic reports placed in the medical record or sent to their primary care pediatrician
5. Parents refuse consent

Max Age: 28 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: The study population will be recruited from Hospital inpatient population, primarily the neonatal intensive care unit who has some anomaly or abnormal laboratory testing suggestive of a genetic disease.
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2015-10-01 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Mortality | At corrected age of 18 months
  The relative frequency of deaths in each group.
Disability Rate | At corrected age of 18 months
  Disability, defined as a physical or mental handicap, especially one that prevents a person from living a full, normal life or from holding a gainful job.
Gene Mutation | In 30 days after receipt of the sample
  To detect the mutation and characterize the genetic architecture and risk variants of neonatal malformation using different genomic methods.

SECONDARY OUTCOMES:
Neurodevelopment(Bayley Scores) | At corrected age of 18 months
  To evaluate neurodevelopmental function by Bayley Scores of Infant Development Mental Development Index (MDI), gain Incidence of MDI<70(Severe) or MDI<85(Moderate)
Respiratory Support | In 14 days after results disclosure
  To observe whether the clinical mornitoring will be changed after results disclosure
Care Level | In 14 days after results disclosure
  To observe whether the care level will be changed after results disclosure

OTHER OUTCOMES:
The total cost for hospitalization | At corrected age of 18 months
  Determination of utilization of healthcare resources in hospital charges in both arms.
Average days of hospitalization | At corrected age of 18 months
  From hospital to discharge.
Parents' understanding of study results | At corrected age of 3 months
  Assessed in parent surveys via questions assessing: subjective understanding, importance of understanding.
Parents' recall of study results | At corrected age of 3 months
  Assessed in parent surveys via questions assessing: results recall

CONTACTS AND LOCATIONS:
Overall Officials: Wenhao Zhou, Doctor, Study Chair — Children's Hospital of Fudan University
Locations (1):
- Children Hospital of Fudan University, Shanghai, Shanghai Municipality, China

REFERENCES:
- [Background] Viggiano E, Marabotti A, Burlina AP, Cazzorla C, D'Apice MR, Giordano L, Fasan I, Novelli G, Facchiano A, Burlina AB. Clinical and molecular spectra in galactosemic patients from neonatal screening in northeastern Italy: structural and functional characterization of new variations in the galactose-1-phosphate uridyltransferase (GALT) gene. Gene. 2015 Apr 1;559(2):112-8. doi: 10.1016/j.gene.2015.01.013. Epub 2015 Jan 13. PMID 25592817
- [Background] Yang D, Sun YY, Bhaumik SK, Li Y, Baumann JM, Lin X, Zhang Y, Lin SH, Dunn RS, Liu CY, Shie FS, Lee YH, Wills-Karp M, Chougnet CA, Kallapur SG, Lewkowich IP, Lindquist DM, Murali-Krishna K, Kuan CY. Blocking lymphocyte trafficking with FTY720 prevents inflammation-sensitized hypoxic-ischemic brain injury in newborns. J Neurosci. 2014 Dec 3;34(49):16467-81. doi: 10.1523/JNEUROSCI.2582-14.2014. PMID 25471584
- [Background] Scully MA, Farrell PM, Ciafaloni E, Griggs RC, Kwon JM. Cystic fibrosis newborn screening: a model for neuromuscular disease screening? Ann Neurol. 2015 Feb;77(2):189-97. doi: 10.1002/ana.24316. Epub 2014 Dec 13. PMID 25425541
- [Background] Hamilton ST, van Zuylen W, Shand A, Scott GM, Naing Z, Hall B, Craig ME, Rawlinson WD. Prevention of congenital cytomegalovirus complications by maternal and neonatal treatments: a systematic review. Rev Med Virol. 2014 Nov;24(6):420-33. doi: 10.1002/rmv.1814. Epub 2014 Oct 14. PMID 25316174
- [Background] Matic M, Simons SH, van Lingen RA, van Rosmalen J, Elens L, de Wildt SN, Tibboel D, van Schaik RH. Rescue morphine in mechanically ventilated newborns associated with combined OPRM1 and COMT genotype. Pharmacogenomics. 2014 Jul;15(10):1287-95. doi: 10.2217/pgs.14.100. PMID 25155931
- [Background] Kwan A, Abraham RS, Currier R, Brower A, Andruszewski K, Abbott JK, Baker M, Ballow M, Bartoshesky LE, Bonilla FA, Brokopp C, Brooks E, Caggana M, Celestin J, Church JA, Comeau AM, Connelly JA, Cowan MJ, Cunningham-Rundles C, Dasu T, Dave N, De La Morena MT, Duffner U, Fong CT, Forbes L, Freedenberg D, Gelfand EW, Hale JE, Hanson IC, Hay BN, Hu D, Infante A, Johnson D, Kapoor N, Kay DM, Kohn DB, Lee R, Lehman H, Lin Z, Lorey F, Abdel-Mageed A, Manning A, McGhee S, Moore TB, Naides SJ, Notarangelo LD, Orange JS, Pai SY, Porteus M, Rodriguez R, Romberg N, Routes J, Ruehle M, Rubenstein A, Saavedra-Matiz CA, Scott G, Scott PM, Secord E, Seroogy C, Shearer WT, Siegel S, Silvers SK, Stiehm ER, Sugerman RW, Sullivan JL, Tanksley S, Tierce ML 4th, Verbsky J, Vogel B, Walker R, Walkovich K, Walter JE, Wasserman RL, Watson MS, Weinberg GA, Weiner LB, Wood H, Yates AB, Puck JM, Bonagura VR. Newborn screening for severe combined immunodeficiency in 11 screening programs in the United States. JAMA. 2014 Aug 20;312(7):729-38. doi: 10.1001/jama.2014.9132. PMID 25138334
- [Background] Morrone A, Caciotti A, Atwood R, Davidson K, Du C, Francis-Lyon P, Harmatz P, Mealiffe M, Mooney S, Oron TR, Ryles A, Zawadzki KA, Miller N. Morquio A syndrome-associated mutations: a review of alterations in the GALNS gene and a new locus-specific database. Hum Mutat. 2014 Nov;35(11):1271-9. doi: 10.1002/humu.22635. Epub 2014 Sep 17. PMID 25137622
- [Background] Mercimek-Mahmutoglu S, Cordeiro D, Cruz V, Hyland K, Struys EA, Kyriakopoulou L, Mamak E. Novel therapy for pyridoxine dependent epilepsy due to ALDH7A1 genetic defect: L-arginine supplementation alternative to lysine-restricted diet. Eur J Paediatr Neurol. 2014 Nov;18(6):741-6. doi: 10.1016/j.ejpn.2014.07.001. Epub 2014 Jul 27. PMID 25127453
- [Background] Eldar-Geva T, Srebnik N, Altarescu G, Varshaver I, Brooks B, Levy-Lahad E, Bromiker R, Schimmel MS. Neonatal outcome after preimplantation genetic diagnosis. Fertil Steril. 2014 Oct;102(4):1016-21. doi: 10.1016/j.fertnstert.2014.06.023. Epub 2014 Jul 23. PMID 25064409
- [Derived] Chen X, Yan K, Gao Y, Wang H, Chen G, Wu B, Qin Q, Yang L, Zhou W. Feeding difficulty is the dominant feature in 12 Chinese newborns with CHD7 pathogenic variants. BMC Med Genet. 2019 May 30;20(1):93. doi: 10.1186/s12881-019-0813-z. PMID 31146700
- See also: Surveying Parents About Genome Screening of Newborns — http://ClinicalTrials.gov/show/NCT01736501
- See also: Gene Therapy for Netherton Syndrome — http://ClinicalTrials.gov/show/NCT01545323
- See also: Genes Associated With Bronchopulmonary Dysplasia and Retinopathy of Prematurity — http://ClinicalTrials.gov/show/NCT01780155
- See also: Clinical Characteristics and Genetic Profiles of Severe Combined Immunodeficiency in China — http://ClinicalTrials.gov/show/NCT02231983
- See also: Gene Transfer for X-Linked Severe Combined Immunodeficiency in Newly Diagnosed Infants — http://ClinicalTrials.gov/show/NCT01512888